CLINICAL TRIAL: NCT04320381
Title: Qualitative Understanding of Experiences With the SIMPLIFY Trial
Acronym: QUEST
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Gregory Sawicki, Co-Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-P00034269; STRC-113-20-01 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis; Drug Withdrawal
Keywords: qualitative; treatment withdrawal
MeSH Terms: conditions — Cystic Fibrosis; Substance Withdrawal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A: subjects in the hypertonic saline study randomized to discontinue or maintain therapy
  Interventions: Behavioral: Qualitative Interview
- Group B: subjects in the dornase alfa study randomized to discontinue or maintain therapy
  Interventions: Behavioral: Qualitative Interview
- Group C: subjects who were randomized but withdrew early from the SIMPLIFY Study.
  Interventions: Behavioral: Qualitative Interview
- Group D: subjects in the hypertonic saline study randomized to discontinue or maintain therapy with FEV1% predicted between 40 and <60%
  Interventions: Behavioral: Qualitative Interview
- Group E: caregiver participants (parents and legal guardians of eligible patient participants less than 18 years of age who were randomized in the SIMPLIFY study)
  Interventions: Behavioral: Qualitative Interview

INTERVENTIONS:
Behavioral: Qualitative Interview — 2 Semi-Structured Qualitative Interviews

SUMMARY:
This qualitative longitudinal study is designed to elicit and thematically analyze the perspectives of SIMPLIFY subjects about treatment withdrawal research and treatment burden in the context of triple combination CFTR (Cystic Fibrosis Transmembrane Conductance Regulator) modulator therapy (TCT). Cohorts will be determined based on sub-groups of the assigned treatment arms from the SIMPLIFY study. Participants will be asked to participate in two interviews; the first interview will be conducted at the completion of the SIMPLIFY study and the second interview will be conducted approximately 4 months after the first interview. Trained research staff will conduct the semi-structured interviews that will be audio-recorded and transcribed for thematic analysis. Each interview should last between 30-60 minutes.

DETAILED DESCRIPTION:
The recommended daily treatment regimen for CF is complex and results in high treatment burden for many people with CF (PwCF). Newly developed triple combination CFTR modulator therapy (TCT) has shown dramatic health benefits on top of standard CF therapies in a pivotal clinical trial and will soon be a treatment option for a larger population of PwCF. Widespread implementation of TCT will provide an unprecedented opportunity to rigorously study whether PwCF can safely discontinue some previously prescribed daily therapies. The randomized, open-label SIMPLIFY study has been designed to test the hypothesis that withdrawal of dornase alpha and/or nebulized hypertonic saline (HS) is not inferior to continuation of one or both treatments with respect to short-term change in lung function. As this is the first of its kind study design in CF, it unknown how people with CF thinking about withdrawal studies or discontinuing treatments.

Here, the investigators intend to conduct a qualitative interview study that complements the SIMPLIFY protocol in which the investigators aim to assess the experiences of PwCF participating in a treatment withdrawal study. In particular, the investigators will examine post-hoc the beliefs and opinions of a representative subgroup of SIMPLIFY participants about treatment withdrawal research and perceived treatment burden. This qualitative study will provide the opportunity to learn about behaviors after the SIMPLIFY trial, including restarting vs. continuing to maintain medications, withdrawing other medications or therapies, and how patients and families partner with care teams around these decisions. Through these interviews, the investigators will learn how individuals with CF perceive taking part in a drug withdrawal study and how participants discern treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

Patient Participant:

1. Participant was randomized into the SIMPLIFY study
2. Person with CF is ≥ 14 years of age at the time of randomization into SIMPLIFY
3. Is English speaking
4. Participant has provided consent (or assent if applicable) in the SIMPLIFY study to provide contact information and share data from the SIMPLIFY study with the QUEST study team
5. Participant has provided contact information via the QUEST portal
6. Is willing and able to adhere to the study requirements
7. Provides consent (or assent if applicable) for the QUEST study
8. Completed participation in the SIMPLIFY study (i.e. completed through Visit 3 or early withdrawal, if applicable)

Caregiver Participant:

1. Lives in the same household as a child with CF who is ≥ 14 years of age but <18 years of age who meets the eligibility requirements for the QUEST study
2. Is English speaking,
3. Is willing and able to adhere to the study requirements
4. Provides consent for the QUEST study

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any situation that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient participants will consist of male and female Cystic Fibrosis patients ages 14 and older who were randomized in the SIMPLIFY study. QUEST researchers will focus on assuring a balanced distribution across sub-groups (see "Groups and Interventions" section for sub-group descriptions).
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Interview #1 | to be conducted at the time of enrollment (post SIMPLIFY study)
  Questions to evaluate (A) attitudes and beliefs regarding participation in a withdrawal study and (B) perceptions of treatment burden in the context of having participated in a withdrawal study.
Interview #2 | to be conducted 4 months following the date of the first interview
  Questions to evaluate pwCF's perceptions of (A) factors that affected the decision to use or not use dornase alfa and/or hypertonic saline post-trial participation and satisfaction with the decision and (B) factors that would affect decision-making about whether to withdraw treatments in the future.

SECONDARY OUTCOMES:
Change in Participant's Perceptions in Interviews | from day one to approximately month 8
  To determine if perceptions about treatment burden and withdrawal study participation vary by the parent study treatment arm assignment (e.g. randomized to continue or stop dornase alfa and/or hypertonic saline).
Change in Participant's Decision-making in Interviews | from day one to approximately month 8
  To determine if treatment arm assignment influenced decision-making about using or not using dornase alfa and/or hypertonic saline post-trial participation
Change in Participant's Level of Satisfaction in Interviews | from day one to approximately month 8
  To determine pwCF's level of satisfaction with the decision to use or not use dornase alfa and/or hypertonic saline post-trial participation

OTHER OUTCOMES:
Change in Participant Perceptions | from day one to approximately month 8
  To determine if individuals who did not maintain treatment assignment (i.e., person randomized to discontinue treatment restarted the treatment OR person randomized to maintain treatment discontinued it) have different perceptions about treatment burden
Change in Participant Perceptions (2) | from day one to approximately month 8
  To determine if individuals who withdrew from the SIMPLIFY study have a different perception about treatment burden and the factors that affect decisions to discontinue treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sawicki, MD, MPH, Principal Investigator — Boston Children's Hospital; Kristin Riekert, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang C, Montgomery M. Dornase alfa for cystic fibrosis. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD001127. doi: 10.1002/14651858.CD001127.pub5. PMID 33735508